CLINICAL TRIAL: NCT06727240
Title: A Non-Inferiority Randomized Clinical Trial Investigating Efficacy and Safety of an Innovative Medical Device in the Reduction of Mechanical Complications of Peripheral Intravenous Catheters
Brief Title: Safe-Infusion Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Interlinked AB (Industry)
Collaborators: Parc Sanitari Sant Joan de Déu (Other); Unidade Local de Saúde de Coimbra, EPE (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Interlinked 05-01-11
Record Dates: First submitted 2024-11-29; First posted 2024-12-10 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Intravenous Access; Medical Device
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ReLink® (Experimental): One or more investigational devices will be added to the infusion line. Standard practise procedure related to PIVC infusions according to hospital norm will be followed. Thereafter the planned IV therapy is initiated until completion.
  Interventions: Device: Intervention
- Control (No Intervention): Standard practise related to PIVC infusions according to hospital norm will be followed. Thereafter the planned IV therapy is initiated until completion.

INTERVENTIONS:
Device: Intervention — The interventional device is a coupling device intended to prevent mechanical complications during peripheral intravenous infusions. While control will not receive the device.
  Arms: ReLink®

SUMMARY:
Around 1.5 billion peripheral intravenous catheters (PIVCs) are sold yearly, with up to 90% of hospitalized patients receiving one, yet failure rates can reach 69%, often due to phlebitis, infiltration, occlusion, or dislodgement. These complications can collectively be named mechanical complications. This study aims to assess a new device's effectiveness in reducing mechanical complications associated with PIVCs through a non-inferiority randomized trial at two sites. A total of 548 patients will be recruited, with primary outcomes focused on complication rates and secondary outcomes examining adverse events, healthcare feedback, and economic impacts.

DETAILED DESCRIPTION:
It is estimated that around 1.5 billion PIVC are sold yearly throughout the globe, and placing them is one of the most common invasive procedures in hospitalised patients, with up to 90% receiving one, yet there is a failure rate of up to 69%.1-5 Some of the most common causes of failure are considered to be phlebitis, subcutaneous infiltration, occlusion and dislodgement. These failure rates vary widely throughout the globe, where published data suggests rates of 8-44% for phlebitis, 5-21% for infiltration, 7.6-16% for occlusion and 5-10% for dislodgement.4,6-12 Phlebitis, commonly defined as an inflammatory process in the wall of a vein, resulting in a blood clot formation; while infiltration is defined as the inadvertent leakage of a solution into the surrounding tissue; occlusion is defined as catheter failure due to blockage, and dislodgement the accidental/ in adverted removal of the PIVC before intended.13 Previous studies have suggested that mechanical irritation could be an important factor resulting in PIVC failure.14-16 In the case of phlebitis, mechanical movements against the endothelial wall could initiate a cascade of prothrombotic events resulting in the formation of a blood clot, something that has been demonstrated in a simulated environment.14,17,18 Furthermore micromechanical movements of the PIVC could eventually lead the PIVC to migrate from within the vessel wall to be unintentionally placed outside the vessel, yet, still in the surrounding tissue causing infiltration. Occlusion is the sudden block of the PIVC, where flushing or aspirating from the PIVC is not possible. Dislodgement of a PIVC is the act of mechanical movement of the PIVC from the intravascular space to the surrounding environment outside of the body.

Therefore, there is a need to investigate potential new methods for prevention of these mechanical complications, and one method could be in the reduction of mechanical forces acting on the vessels. The aim of this study is to investigate the safety and effectiveness of a new medical device in reducing the number of mechanical complications during IV therapy.

To answer this aim, a non-inferiority randomized clinical trial will be executed at two sites, where patients having a vascular access will be examined in a systematic fashion. Inclusion criteria are: having VAD, >18 years of age, speak local language, absence of signs of phlebitis or infiltration, and a signed consent form. Exclusion criteria are: VAD for sampling only, pregnancy, unable to obtain informed consent, patients under palliative care and VAD for bolus infusion only.

A total of 548 patients will be recruited to this study, and it is estimated to take 5 months to complete. The primary outcomes/endpoints are to investigate the rate of mechanical complications in the form of phlebitis, infiltration, occlusion and dislodgement. While secondary outcomes/endpoints will be identifying the frequency and severity of any adverse events, healthcare opinions on the device and the economic burden of the mechanical complications. No follow up is planned in this trial.

ELIGIBILITY:
Inclusion Criteria:

* The patient has or will get a vascular access device (VAD) expected to be used for continuous or intermittent IV infusion therapy. Continuous IV infusion is defined as an infusion ≥2h and intermitted as an infusion lasting 15min to <2h.
* ≥18 years of age
* Speak and understand local language
* VADs already in place when the patient is admitted to the ward should not present with phlebitis or infiltration or occlusion
* Participants have signed the informed consent or have a legal authorized representative (LAR) who has provided this consent

Exclusion Criteria:

* The VAD is expected to be used for sampling only
* Pregnancy
* Unable to obtain informed consent or without an available LAR to provide surrogate informed consent
* Patients under palliative care
* Bolus IV infusion, defined as an infusion time of <15 min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 548 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
The rate of mechanical complications of an IV therapy session using the device compared to using current 'state of the art'. | Baseline PIVC data and immediatly after PIVC removal
  Mechanical complications are defied as following:
  * Phlebitis -inflammation of a vein based on clinical diagnosis
  * Infiltration - the process of accidental leakage of fluids out of the veins into peripheral tissue
  * Occlusion - blocked PIVC, where flushing or aspirating from the PIVC is not possible
  * Dislodgment - the process of accidental/ unintentional complete removal of the PIVC before scheduled removal

SECONDARY OUTCOMES:
Frequency and severity of any adverse events | Through study participation (hospitlized in the ward), an average of 5 days
Healthcare workers opinion of investigational device | Immediately after the intervention
  A questionnaire has been developed asking baseline data from healthcare worker. The questionnaire contains questions about 1) opinion about using the device again, 2) recommendation of the device, and 3) usage of the device for a relative. Each question is ranked from 0 to 5.
The economic cost of these disruptions to your facility in terms of man-hours, and resources. | Immediatly after PIVC removal

CONTACTS AND LOCATIONS:
Overall Officials: Ramon Mir Abellán, PhD, Principal Investigator — Parc Sanitari Sant Joan de Déu; António Manuel Marques, PhD, Principal Investigator — Unidade Local de Saúde de Coimbra, EPE
Locations (2):
- Centro Hospitalar e Universitário de Coimbra, Coimbra, Portugal
- Parc Sanitari Sant Joan de Déu, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
All research results will be reported at a de-identified level, and any statistical correlations linked to personal data in terms of gender and/or age will be reported at an aggregated level.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 1 year of study completion